CLINICAL TRIAL: NCT02219893
Title: Phase I/II Trial of MOC31PE Immunotoxin in Peritoneal Carcinomatosis From Colorectal Carcinoma
Brief Title: Immunotoxin in Peritoneal Carcinomatosis- ImmunoPeCa Trial
Acronym: ImmunoPeCa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, Senior consultant medical oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ImmunoPeCa Trial
Record Dates: First submitted 2014-08-08; First posted 2014-08-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Neoplasms
Keywords: Peritoneal Carcinomatosis; Peritoneal Metastasis; Colorectal Cancer; Cytoreductive surgery; HIPEC; Intraperitoneal treatment; Immunotoxin; MOC31PE
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — MOC31PE immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MOC31PE Immunotoxin (Experimental): Drug to be instilled on day 1 after cytoreductive surgery and HIPEC.
  Interventions: Drug: MOC31PE Immunotoxin

INTERVENTIONS:
Drug: MOC31PE Immunotoxin — Patients who meet inclusion criteria will be treated with a single intraperitoneal MOC31PE immunotoxin instillation for 6 hours on the first day after CRS and HIPEC

SUMMARY:
The purpose of this study is through a phase I/II clinical trial to assess the safety and toxicity of intraperitoneally administered MOC31PE immunotoxin, given on the 1.postoperative day after cytoreductive surgery (CRS) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for peritoneal metastases from colorectal cancer (CRC).

DETAILED DESCRIPTION:
MOC31PE is an immunotoxin that has previously been evaluated in a phase I clinical study involving patients with advanced EpCAM positive carcinoma to assess the safety and tolerability profile and the pharmacokinetic behavior of the compound. In this study, the compound was administered intravenously and was well tolerated. MOC31PE will now be evaluated on the same parameters in a new phase I/II clinical trial, where the drug will be administered intraperitoneally to patients with peritoneal metastases from EpCAM positive colorectal carcinomas.

ELIGIBILITY:
Inclusion criteria:

* Histologically verified EpCAM positive colorectal cancer
* Ambulatory with Eastern Cooperative Oncology Group (ECOG) performance status 0-1 at the time of surgery
* At least 18 years of age
* Suspected isolated peritoneal carcinomatosis upon radiologic work-up
* Complete cytoreduction at surgery and mitomycin C given as standard HIPEC procedure
* Peritoneal Cancer Index (PCI) ≤ 20
* Laboratory values at inclusion:

  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  * Platelets > 100 x 10^9/L
  * Hb > 9g/dL
  * Creatinine ≤ 2x upper limit of normal
  * Bilirubin < 2.0x the upper limit of normal
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2. 5x the upper limit of normal
  * Albumin levels > 30 g/L
  * International normalised ratio (INR) <1.3
* Signed informed consent and expected cooperation with respect to treatment and follow-up must be obtained and documented according to International Conference of Harmonisation- Good clinical Practice (ICH GCP), and national/local regulations.

Exclusion criteria:

* Other synchronous metastatic lesions. Patients may be included if they have had curative resection of metastatic CRC disease more than 2 years prior to inclusion and have no relapse at this location is detected.
* History of prior other malignant disease the last 3 years, except for adequately treated carcinoma of the cervix or basal or squamous cell skin cancer.
* History of central nervous system (CNS)- or bone metastases
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* History of any liver disease including Hepatitis B or C infection
* Chemotherapy/radiation therapy or major surgery within the last 4 weeks before start of treatment
* BMI > 35
* Pregnant or breast-feeding patients
* Alcohol or drug abuse
* Use of drugs that can influence hepatic function (e.g. phenytoin or phenobarbital)
* Use of anticoagulants
* Any reason why, in the opinion of the investigator, the patient should not participate in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 years or until disease progression
  Follow-up: 5 years from administration of study drug, or until disease progression

SECONDARY OUTCOMES:
Cmax, Tmax | 8 weeks
  Measurements will be done at 0, 3, 6, 12, 24, 48 and 72 hours after administration of study drug
Neutralizing anti-immunotoxin antibody response | 8 weeks
  Measurements of neutralizing anti-immunotoxin antibody response will be done at 4 and 8 weeks after administration of study drug
Biomarkers of disease recurrence | 5 years or until disease progression
  Serum samples for identification of biomarkers of disease recurrence will be taken at every follow-up for 5 years or until disease progression
Overall survival | 5 years
  Overall survival of all patients will be assessed after 5 years
Disease free survival | 5 years
  Follow up period of 5 years, or until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Flatmark, MD PhD, Principal Investigator — Oslo University Hospital; Svein Dueland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital- The Norwegian Radium Hospital, Oslo, Norway